CLINICAL TRIAL: NCT00775476
Title: Treatment of Systemic Lupus Erythematosus (SLE) With N-acetylcysteine (NAC) (SNAC)
Brief Title: Treatment of Systemic Lupus Erythematosus (SLE) With N-acetylcysteine
Acronym: NAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Cedars-Sinai Medical Center (Other); University of Rochester (Other); Yale University (Other); Penn State University (Other); Hospital for Special Surgery, New York (Other); Ohio State University (Other); Oklahoma City VA Health Care System (U.S. Federal Agency); St. Luke's Hospital and Health Network, Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRBnet # 1566736; NIH Award #1U01AR076092 - 01A1
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus (SLE), an autoimmune disease
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: This study will titrate to tolerance during an initial 3 month open label period and then subjects will be randomized to one of 2 arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NAC (Active Comparator): 2.4 g - 4.8 g of NAC daily starting after 3 month open label titration period.
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): 2.4 g - 4.8 g of placebo per day after 3 month open label titration period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — Capsules of NAC, each containing 600 mg of NAC between dosages of 2.4 g to 4.8 g daily
  Arms: NAC
Drug: Placebo — placebo (sugar) twice daily, daily dosage will match that of NAC that was tolerated between daily dosages of 2.4 g and 4.8 g during the open-label titration phase.
  Arms: Placebo

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic inflammatory disease which often has debilitating and potentially life-threatening consequences. The cause of SLE is unknown and current therapies lack specificity and carry significant side-effects. We previously discovered the depletion of glutathione in lymphocytes of patients with SLE and associated this metabolic change with the elevation of the mitochondrial transmembrane potential.

This study will titrate to tolerance during an initial 3 month open label period and then subjects will be randomized to one of 2 arms.

It was determined by statistical analysis that each group must have 105 subjects. All subjects will be enrolled and evaluated for tolerance of NAC between dosages of 2.4 g/day and 4.8 g/day for 3 months. After A 3-month open-label dose-titration phase, SLE subjects will be randomized into 2 groups of 105 subjects either to continue the tolerated dosage of NAC or switched to equal number of placebo capsules. There will be up to seven study visits per SLE subject, including the screening and wash out visits. Visits 2-6 will be scheduled three months apart. The study will last 13 months with the wash-out visit. Each subject will donate approximately 100 ml of blood for biomarker studies at each visit. Healthy control subjects will donate blood at the same time. They will be matched to the SLE subjects by gender, age within 10 years, and ethnicity. Their blood will be used as reference for biomarker assays.

There is a consent form required to participate in the phase II study.

DETAILED DESCRIPTION:
Subjects will take NAC in a dose range of 2.4 g/day to 4.8 g/day which will be titrated to tolerance during an initial 3-month open label period. After the 3-month open label period, patients in each arm will continue taking equal numbers of capsules representing a dosage that has been titrated to tolerance. As an example, the patients tolerating 2.4 g/day, or 4 capsules containing 600 mg of NAC, after 3 months will be randomized to take 4 NAC or 4 placebo (2.4 g/day dextrose) capsules twice daily for the 9 subsequent months.

The primary outcome variable will be the response (yes/no) in the SLE Respinder Index or SRI at Month 12 (reduction ≥ 4 points in SELENA-SLEDAI score and therefore also called SRI-4; no new BILAG A organ domain score and no more than 1 new BILAG B organ domain score; and no worsening in Physician's Global Assessment (PGA) score) by ≥ 0.3 points versus baseline). A positive response will also require no treatment failure, defined as the need for non-protocol treatment, i.e., new or increased immunosuppressives or antimalarials; increased or parenteral corticosteroids; or premature discontinuation from study treatment. Corticosteroids can be tapered off at the investigator's discretion, based on disease activity. Four weeks after randomization, once tapered, corticosteroids can only be increased again to the dosage preceding the last taper step; any larger increase will be deemed a treatment failure. In addition, any increase in corticosteroid dosage during the last 3 months of the trial will result in declaration of treatment failure.

We will monitor tolerance and safety, and assess SLEDAI, BILAG, FAS, PROMIS, ASRS, prednisone use, liver and bone marrow function as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18;
* Male or female;
* ≥ 4 ACR SLE classification criteria (104,105);
* Positive ANA at a titer of ≥ 1/80;
* Stable immunosuppressants (MMF ≤ 3 g/day, azathioprine ≤ 150 mg/day; methotrexate ≤ 25 mg/week; leflunomide ≤ 20 mg/week; cyclosporin 100 mg/day; voclosporin 47.4 mg/day) and/or antimalarials (hydroxychloroquine ≤ 400 mg/day) for 30 days prior to screening; stable oral corticosteroids for 2 weeks prior to screening; ≤ 20 mg/day prednisone or equivalent; stable belimumab or anifrolumab for 90 days prior to screening;
* BILAG 2004 index (48) level A disease activity in ≥ 1 organ/system except renal or central nervous system or BILAG 2004 index level B disease activity in ≥ 1 organs/systems if no level A disease activity is present and SLEDAI ≥ 6 (106);
* Enrollment is approved by adjudication committee within 10 days, which may include retesting and communication with study sites, as necessary.
* Patients may be considered for enrollment 12 months after rituximab treatment, or 6 months after rituximab treatment if their B cell counts have normalized.

Participant Exclusion Criteria

* Acute SLE flare threatening vital organs;
* Pregnant or lactating;
* Moderately serious or serious comorbidities (e.g., diabetes mellitus, congestive heart failure, chronic obstructive pulmonary disease, chronic renal insufficiency) that in investigator's opinion confers high risk for adverse events;
* Patients receiving cyclophosphamide within 3 months;
* Active chronic infections (e.g., HIV, hepatitis B virus, hepatitis C virus, mycobacteria); patients with oral steroid-dependent asthma;
* Infections requiring intravenous antibiotics within a month or oral antibiotics within two weeks of screening; Patients taking (unwilling or unable to stop) NAC or other antioxidants within 1 month of screening (which is considered sufficient time to revert GSH to pre-treatment levels (29);
* Patients who participated in the pilot RCT or are taking daily acetaminophen (≤ 1 g/day prn is allowed if documented);
* Patients receiving mTOR inhibitors (rapamycin/sirolimus, everolimus);
* Patients enrolled in other interventional trials.
* Patients should not take medications containing acetaminophen (Tylenol) as it may reduce the effectiveness of NAC. 1 g/day of acetaminophen is allowed if documented.
* Patients should avoid taking more than 500 mg of vitamin C and more than 30 IU of vitamin E daily as both vitamin C and E can confound the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Therapeutic benefit | 12 months
  Positive response on the SLE Responder Index (SRI) in the NAC arm vs placebo
Improvement of disease activity | 12 months
  Improvement of disease activity as measurable by the reduction of SLEDAI or BILAG disease activity scores and the reduction of prednisone usage
Tolerance and safety | 12 months
  Monitor adverse events and tolerance of the study drug

SECONDARY OUTCOMES:
Immunobiological outcomes measurable improved lymphocyte function | 12 months
  Immunobiological outcomes measurable by improved markers of glutathioen depletion, mitochondrial function and activation of T and B lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Andras Perl, M.D., Ph.D., Principal Investigator — State University of New York - Upstate Medical University
Locations (8):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - Hospital for Special Surgery, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - The Ohio State University, Columbus, Ohio
  - VA Medical Center, Oklahoma City, Oklahoma
  - St. Luke's University Health Network, Allentown, Pennsylvania
  - Penn State MS Hershey Medical Center, Hershey, Pennsylvania

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Lai ZW, Hanczko R, Bonilla E, Caza TN, Clair B, Bartos A, Miklossy G, Jimah J, Doherty E, Tily H, Francis L, Garcia R, Dawood M, Yu J, Ramos I, Coman I, Faraone SV, Phillips PE, Perl A. N-acetylcysteine reduces disease activity by blocking mammalian target of rapamycin in T cells from systemic lupus erythematosus patients: a randomized, double-blind, placebo-controlled trial. Arthritis Rheum. 2012 Sep;64(9):2937-46. doi: 10.1002/art.34502. PMID 22549432